CLINICAL TRIAL: NCT01517100
Title: The Roles of Endocannabinoids in Insulin Secretion and Action
Brief Title: The Role of Endocannabinoids in Insulin Production and Action
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 999912018; 12-AG-N018
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2025-06-10

CONDITIONS: Healthy Volunteers
Keywords: Glucose; Insulin Secretion; Insulin Action; Endocannabinoids; Insulin; Metabolism
MeSH Terms: conditions — Insulin Resistance | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Other: Nabilone — CB agonist
Drug: CP-945,598 — Cannabinoid Receptor 1 antagonist
Other: hyperglycemic clamp — assesses beta cell response
Other: euglycemic-hyperinsulinemic clamp — measures insulin sensitivity
Other: Nabilone — cannabinoid receptor agonist

SUMMARY:
Background:

- The endocannabinoid system is involved in different body functions and processes. It helps regulate appetite and mood, and sends signals to the nervous system. It may also be involved in how the body produces insulin during digestion. Researchers want to test two drugs that work on the endocannabinoid system: nabilone and CP-945,598. These drugs may be able to affect insulin levels in the blood. This information may suggest possible new treatments for people with diabetes.

Objectives:

- To study how the endocannabinoid system is involved in insulin production and action.

Eligibility:

- Healthy men between 21 and 55 years of age.

Design:

* Participants will be screened with a physical exam and medical history. They will provide blood and urine samples. They will also have imaging studies to test their brain responses, especially to food-related cues. Some participants will also have a study visit to test their insulin resistance levels.
* Participants will have four separate study visits 6 weeks apart. They will keep a food diary before each visit. At each visit, they will have one of the following combinations of drugs:
* Double placebo
* Placebo and nabilone
* Placebo and low dose of CP-945,598
* Placebo and high dose of CP-945,598.
* Participants will have follow-up visits 1 week after each study visit. Blood samples will be taken.

DETAILED DESCRIPTION:
Objectives and Specific Aims:

We plan to investigate whether the endocannabinoid system is involved in the regulation of insulin secretion from Beta cells and in the modulation of insulin action in peripheral tissues in humans. We hypothesize that cannabinoid receptor 1 (CB1R) antagonist CP-945,598 will increase insulin secretion from Beta cells and improve insulin sensitivity in peripheral tissues while cannabinoid receptor (CBR) agonist nabilone will decrease insulin secretion from Beta cells and worsen insulin sensitivity in peripheral tissues. Moreover, we will investigate the brain s control over the initial phase of insulin secretion (cephalic insulin response) and the effect of central cannabinoid receptors.

Experimental Design and Methods:

Twenty healthy men, age 21-55, will be recruited for this study. This is a randomized, double-blind, placebo-controlled cross-over study. Each subject will serve as his own control and each person will have four different intervention visits spaced at least 6 weeks apart. During each visit, they will receive one of the following medications in random order: placebo, nabilone 2 mg, CP-945,598 15 mg, or CP-945,598 45 mg. A sequential hyperglycemic-euglycemic clamp procedure and a 3-hr oral glucose tolerance test will be used to study the effect of CP-945,598 and nabilone on insulin secretion and insulin action in healthy men. To identify brain areas involved in cephalic insulin response, a functional MRI will be used to assess brain activation in response to food images in association with frequent blood sampling.

Medical Relevance and Expected Outcome:

Based on our pre-clinical animal data, CB1R antagonist enhances insulin secretion and action in response to glucose while CBR agonist virtually shuts off insulin secretion and worsens insulin action in response to glucose. The application of novel, pre-clinical findings to an understanding of human biology and pathobiology is of fundamental and critical importance. This study will give us a better understanding of the regulators of insulin secretion from Beta cells and insulin sensitivity in humans, and this new understanding is of importance to finding new treatments for type 2 diabetes.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Healthy men only

     (We want to study men because the magnitude of acute insulin response for men and women is different. In addition, as women may become pregnant in the course of the study, and since this is a physiology study only, and not one related to treatments, we want to remove any confounders and lessen any chance of drop-out.)
  2. Age 21-55 (Age restriction is used to remove age as a confounding factor because Beta cells function tends to deteriorate and first phase secretion becomes less defined with age.
  3. Screening laboratory evaluations with no clinically significant abnormal results (minor deviations from normal lab results will be at the discretion of the principal investigator):

     1. fasting comprehensive metabolic panel
     2. complete blood count with differential and platelet
     3. thyroid function test (TSH, free T4)
     4. urinalysis
     5. urine drug screen
  4. BMI less than 30 (Men with BMI greater than or equal to 30 are excluded because obesity has been associated with altered beta cell function.
  5. Have NOT participated in another clinical trial involving any pharmacologic agents within the past 30 days
  6. Able to complete an inform consent
  7. Agree to not participate in other clinical trials within the study period (at the discretion of the study investigator)

EXCLUSION CRITERIA:

1. Women
2. FPG greater than or equal to 100 mg/dl or 2-hr OGTT greater than or equal to 140 mg/dL
3. Evidence of illicit drug use
4. History of substance abuse including marijuana within the past 6 months
5. History of smoking any tobacco products within six months prior to screening
6. Alcohol intake greater than 30 grams (drink more than 2 beers per day OR equivalent amount of alcohol)
7. History of Human Immunodeficiency Virus (HIV) infection
8. History of active or chronic Hepatitis B and/or C infection
9. History of malignancy
10. History of coronary disease
11. History of seizures or other neurologic diseases
12. History of psychiatric illnesses including major depressive disorder, schizophrenia, bipolar disorder
13. Any lifetime history of suicide attempt
14. History of suicidal behavior in the last year
15. Any suicidal behavior during any follow-up visits
16. History of any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale

    (C-SSRS) in the last year
17. Any suicidal ideation of type 4 or 5 on the C-SSRS during any follow-up visits.
18. Patient Health Questionnaire-9 (PHQ-9) score greater than or equal to 10 during screening visit or any follow-up study visits
19. Generalized Anxiety Disorder-7 (GAD-7) score greater than or equal to 10 during screening visit or any follow-up visits
20. History of liver or renal diseases
21. History of gastrointestinal or endocrine disorders
22. History of glucocorticoid use (over one month) or other immunosuppressive agents (any)
23. Any condition or non-removable device contraindicated for MRI (pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments, or history of working as a welders or metal worker)
24. Any medical history that, in the opinion of the investigator(s), will make participation of the subject in the study unsafe

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01-05; Primary Completion 2014-10-06 (Actual); Study Completion 2014-10-06 (Actual)

PRIMARY OUTCOMES:
Changes in insulin sensitivity. | CB1R antagonist CP-945,598 will enhance while CR receptor agonist nabilone will suppress first phase insulin response fromB cells in humans
  This study will give us a better understanding of the regulators of insulin secretion from B cells and insulin sensitivity in humans and this new understanding is of importance to finding new treatments for type 2 diabetes

SECONDARY OUTCOMES:
Changes in insulin and other hormones and the brain response to picture of food items evidenced by functional MRI of the brain. | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Chee W Chia, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The NIA IRP is discussing the plan to make IPD available. A final decision has not been made.

REFERENCES:
- [Background] Pratley RE, Weyer C. The role of impaired early insulin secretion in the pathogenesis of Type II diabetes mellitus. Diabetologia. 2001 Aug;44(8):929-45. doi: 10.1007/s001250100580. PMID 11484070
- [Background] Straub SG, Sharp GW. Hypothesis: one rate-limiting step controls the magnitude of both phases of glucose-stimulated insulin secretion. Am J Physiol Cell Physiol. 2004 Sep;287(3):C565-71. doi: 10.1152/ajpcell.00079.2004. PMID 15308461
- [Background] Elahi D, Muller DC, McAloon-Dyke M, Tobin JD, Andres R. The effect of age on insulin response and glucose utilization during four hyperglycemic plateaus. Exp Gerontol. 1993 Jul-Oct;28(4-5):393-409. doi: 10.1016/0531-5565(93)90066-m. PMID 8224037